CLINICAL TRIAL: NCT06205446
Title: Application of Diaphragmatic Breathing in Patients With Disorders of Gut-brain Interaction: Impact on Gastrointestinal and Psychological Symptoms as Well as Autonomic Nervous System
Brief Title: Application of Diaphragmatic Breathing in Patients With Disorders of Gut-brain Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB112-185-A
Record Dates: First submitted 2023-12-28; First posted 2024-01-16 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-08

CONDITIONS: Irritable Bowel Syndrome; Healthy Subjects; Functional Gastrointestinal Disorders; Laryngopharyngeal Reflux
Keywords: Heart rate variability; Diaphragmatic breathing; Gut-brain axis dysregulation
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases; Laryngopharyngeal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- abdominal breathing (Experimental): The relationship between respiration and the autonomic nervous system (ANS) is closely intertwined, as the phrenic nerve, responsible for controlling the movement of the diaphragm, is connected to the vagus nerve of the parasympathetic nervous system.The respiratory cycle reflects the balance between the parasympathetic and sympathetic nervous systems in the Autonomic Nervous System (ANS), which can be observed through Heart Rate Variability (HRV). The ANS state shifts from the parasympathetic nervous system to the sympathetic nervous system during inhalation, while it transitions from the sympathetic nervous system to the parasympathetic nervous system during exhalation. In HRV, an increase in heart rate indicates enhanced sympathetic nervous system activity during inhalation, whereas a decrease in heart rate signifies increased parasympathetic nervous system activity during exhalation.
  Interventions: Behavioral: Healthy subjects : abdominal breathing; Behavioral: Laryngopharyngeal reflux disease subjects : abdominal breathing; Behavioral: Dyspepsia subjects : abdominal breathing; Behavioral: Irritable bowel disorder : abdominal breathing

INTERVENTIONS:
Behavioral: Healthy subjects : abdominal breathing — The guidance content for the second session of self-practice in the first week involves practicing for 5 minutes each day, and recording a week-long diary of diaphragmatic breathing. After the first week, the subjects will undergo a once-off autonomic nervous system test and a questionnaire assessment of physical and mental symptoms. In the second week, the subjects will receive guidance for the second session of daily self-practice, practicing for 5 minutes each time, and recording a week-long diary of diaphragmatic breathing. After the second week, the subjects will undergo another round of autonomic nervous system testing and a questionnaire assessment of physical and mental symptoms.
Behavioral: Laryngopharyngeal reflux disease subjects : abdominal breathing — The guidance content for the second session of self-practice in the first week involves practicing for 5 minutes each day, and recording a week-long diary of diaphragmatic breathing. After the first week, the subjects will undergo a once-off autonomic nervous system test and a questionnaire assessment of physical and mental symptoms. In the second week, the subjects will receive guidance for the second session of daily self-practice, practicing for 5 minutes each time, and recording a week-long diary of diaphragmatic breathing. After the second week, the subjects will undergo another round of autonomic nervous system testing and a questionnaire assessment of physical and mental symptoms.
Behavioral: Dyspepsia subjects : abdominal breathing — The guidance content for the second session of self-practice in the first week involves practicing for 5 minutes each day, and recording a week-long diary of diaphragmatic breathing. After the first week, the subjects will undergo a once-off autonomic nervous system test and a questionnaire assessment of physical and mental symptoms. In the second week, the subjects will receive guidance for the second session of daily self-practice, practicing for 5 minutes each time, and recording a week-long diary of diaphragmatic breathing. After the second week, the subjects will undergo another round of autonomic nervous system testing and a questionnaire assessment of physical and mental symptoms.
Behavioral: Irritable bowel disorder : abdominal breathing — The guidance content for the second session of self-practice in the first week involves practicing for 5 minutes each day, and recording a week-long diary of diaphragmatic breathing. After the first week, the subjects will undergo a once-off autonomic nervous system test and a questionnaire assessment of physical and mental symptoms. In the second week, the subjects will receive guidance for the second session of daily self-practice, practicing for 5 minutes each time, and recording a week-long diary of diaphragmatic breathing. After the second week, the subjects will undergo another round of autonomic nervous system testing and a questionnaire assessment of physical and mental symptoms.

SUMMARY:
Patients with disorders of gut-brain interaction (DGBI) often present gastrointestinal symptoms that do not show noticeable irregularities in standard examinations. However, due to unclear causes and a high prevalence rate, this condition often exerts a profound impact on the physical and mental health of patients. The scope of DGBI encompasses conditions such as laryngopharyngeal reflux, functional dyspepsia, and irritable bowel syndrome. Previous research has confirmed that in patients with DGBI, their autonomic nervous system exhibits an imbalance, charact erized by decreased parasympathetic activity and dominant sympathetic activity. Diaphragmatic breathing helps reduce the respiratory rate and can stimulate parasympathetic activity while suppressing sympathetic activity. Hence, it is now officially recommended as an effective adjunct therapy for relieving symptoms of gastroesophageal reflux. Accordingly, this study plans to implement a randomized controlled trial, introducing diaphragmatic breathing to patients with DGBI who exhibit normal results in objective examinations. This work allows evaluate changes in their psychophysical symptoms before and after treatment, as well as alterations in the autonomic nervous system .

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects:

1. Age between 18 and 70, mentally alert and willing to sign the consent form for the study.
2. No gastrointestinal symptoms or use of gastrointestinal medication.

Inclusion criteria for Laryngopharyngeal reflux disease subjects:

1. Age between 18 and 70, mentally alert and willing to sign the consent form for the study.
2. Gastroesophageal reflux disease (GERD) is defined as the condition characterized by experiencing symptoms for at least three months (such as hoarseness, sensation of a foreign body in the throat, chronic cough, and frequent throat clearing) occurring at least once a week. Reflux Symptom Index (RSI) is a standardized questionnaire for evaluating laryngopharyngeal reflux. It consists of nine reflux-related symptoms, with severity scores ranging from 0 (no symptoms) to 5 (most severe). A total score exceeding 13 indicates the criteria for inclusion of a patient as having laryngopharyngeal reflux.

dyspepsia subjects:

1. Age between 18 and 70, mentally alert and willing to sign the consent form for the study.
2. Those who meet the definition of functional dyspepsia (FD). (Functional dyspepsia is chronic ( once a week , lasting for at least three months, at least six months before the first symptom) upper gastrointestinal symptoms (any of the following ) : postprandial abdominal distension, easy feeling of fullness, upper abdominal pain Or upper abdominal burning sensation, and no symptoms of gastrointestinal bleeding or significant weight loss, no abnormality after upper gastrointestinal endoscopy).

Inclusion criteria for subjects with irritable bowel disorder:

1. Age between 18 and 70, mentally alert and willing to sign the consent form for the study.
2. meet the definition of irritable bowel disorder (IBS) . Irritable bowel syndrome is chronic ( once a week , lasting for at least three months) lower gastrointestinal symptoms: abdominal pain combined with diarrhea or constipation , and no symptoms of gastrointestinal bleeding or significant weight loss, no abnormalities after colonoscopy) .

Exclusion Criteria:

1. Pregnant or lactating women.
2. Infected with antibiotic resistance.
3. Received endotracheal intubation in the past two months .
4. Having myocardial ischemia or recently experienced a myocardial infarction.
5. Unable to collaborate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on the Functional Dyspepsia Scale(FD) at 14 days | Baseline and day 14
  Possible scores range from 0 (Very slightly) to 6 (Very serious) 0=Very slightly 1=Slight 2=A little slightly 3=About medium 4=A bit serious 5=Severe 6=Very serious Change = (day 14 Score - Baseline Score).
Change from Baseline on the Irritable Bowel Syndrome Scale(IBS) at 14 days | Baseline and day 14
  Possible scores range from 1 (Never) to 5 (Always)
  1=Never 2=Sometimes 3=Often4=most of the time 5=Always Change = (day 14 Score - Baseline Score).
Change from Baseline on the Gastroesophageal Reflux Disease Questionnaire(GERDQ) at 14 days | Baseline and day 14
  Possible scores range from 1 (Never) to 3 (4~7days) 0=Never 1=1 day 2=2~3days 3=4~7days Change = (day 14 Score - Baseline Score).
Change from Baseline on the Reflux Symptom Index (RSI) at 14 days | Baseline and day 14
  Possible scores range from 0 (no symptoms) to 5 (most severe) 0= No Problem 1=very slight 2=slight 3=About medium 4=moderate to severe 5=Severe Problem Change = (day 14 Score - Baseline Score).
Change from Baseline in Pain on the Gastrointestinal symptom rating scale (GSRS) at 14 days | Baseline and day 14
  Possible scores range from 1 (No pain) to 4 (Worst possible pain)
  1=No pain 2=Mild 3=Moderate 4=Worst possible pain Change = (day 14 Score - Baseline Score).
Change from Baseline on the Pittsburgh sleep quality index (PSQI) at 14 days | Baseline and day 14
  Possible scores range from 0 (Never) to 3 (Occurs three times a week times or more) 0=Never 1=Less than once a week 2=Occurs once or twice a week 3=Occurs three times a week times or more Change = (day 14 Score - Baseline Score).
Change from Baseline on the Taiwanese Depression Scale (TDQ) at 14 days | Baseline and day 14
  Possible scores range from 0 (Never) to 3 (Always) 0=Never 1=Sometimes 2=Often 3=Always Change = (day 14 Score - Baseline Score).
Change from Baseline on the State-Trait Anxiety Inventory (STAI) at 14 days | Baseline and day 14
  Possible scores range from 1 (Never) to 4 (Always)
  1=Never 2=Sometimes 3=Often 4=Always Change = (day 14 Score - Baseline Score).
Change from Baseline on the Perceived Stress Scale(PSS-10) at 14 days | Baseline and day 14
  Possible scores range from 0 (Never) to 4 (Always) 0=Never 1=Rarely 2=Sometimes 3=Often 4=Always Change = (day 14 Score - Baseline Score).
Change from Baseline on the Esophageal Hypervigilance and Anxiety Scale (EHAS) at 14 days | Baseline and day 14
  Possible scores range from 0 (Strongly disagree) to 4 (Strongly agree) 0=Strongly disagree 1=Somewhat disagree 2=Neiteher agree nor disagree 3=Somewhat agree 4 =Strongly agree Change = (day 14 Score - Baseline Score).
Change from Baseline on the Laryngeal Hypervigilance and Anxiety Scale (LHAS) at 14 days | Baseline and day 14
  Possible scores range from 0 (Strongly disagree) to 4 (Strongly agree) 0=Strongly disagree 1=Somewhat disagree 2=Neiteher agree nor disagree 3=Somewhat agree 4 =Strongly agree Change = (day 14 Score - Baseline Score).
Change from Baseline on the Visceral Sensitivity Index (VSI) at 14 days | Baseline and day 14
  Possible scores range from 1 (Strongly disagree) to 6 (Strongly agree)
  1=Strongly agree 2=Moderately agree 3=Mildly agree 4=Mildly disagree 5 =Moderately disagree 6=Strongly disagree Change = (day 14 Score - Baseline Score).

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Margolis KG, Cryan JF, Mayer EA. The Microbiota-Gut-Brain Axis: From Motility to Mood. Gastroenterology. 2021 Apr;160(5):1486-1501. doi: 10.1053/j.gastro.2020.10.066. Epub 2021 Jan 22. PMID 33493503
- [Result] Drossman DA, Hasler WL. Rome IV-Functional GI Disorders: Disorders of Gut-Brain Interaction. Gastroenterology. 2016 May;150(6):1257-61. doi: 10.1053/j.gastro.2016.03.035. No abstract available. PMID 27147121
- [Result] Wong MW, Hsiao SH, Wang JH, Yi CH, Liu TT, Lei WY, Hung JS, Liang SW, Lin L, Gyawali CP, Chen PR, Chen CL. Esophageal Hypervigilance and Visceral Anxiety Contribute to Symptom Severity of Laryngopharyngeal Reflux. Am J Gastroenterol. 2023 May 1;118(5):786-793. doi: 10.14309/ajg.0000000000002151. Epub 2022 Dec 14. PMID 36693025
- [Result] Drossman DA, Tack J, Ford AC, Szigethy E, Tornblom H, Van Oudenhove L. Neuromodulators for Functional Gastrointestinal Disorders (Disorders of Gut-Brain Interaction): A Rome Foundation Working Team Report. Gastroenterology. 2018 Mar;154(4):1140-1171.e1. doi: 10.1053/j.gastro.2017.11.279. Epub 2017 Dec 22. PMID 29274869
- [Result] Duan H, Cai X, Luan Y, Yang S, Yang J, Dong H, Zeng H, Shao L. Regulation of the Autonomic Nervous System on Intestine. Front Physiol. 2021 Jul 14;12:700129. doi: 10.3389/fphys.2021.700129. eCollection 2021. PMID 34335306
- [Result] Phillips RJ, Powley TL. Innervation of the gastrointestinal tract: patterns of aging. Auton Neurosci. 2007 Oct 30;136(1-2):1-19. doi: 10.1016/j.autneu.2007.04.005. Epub 2007 May 29. PMID 17537681
- [Result] Agusti A, Garcia-Pardo MP, Lopez-Almela I, Campillo I, Maes M, Romani-Perez M, Sanz Y. Interplay Between the Gut-Brain Axis, Obesity and Cognitive Function. Front Neurosci. 2018 Mar 16;12:155. doi: 10.3389/fnins.2018.00155. eCollection 2018. PMID 29615850
- [Result] Callaghan B, Furness JB, Pustovit RV. Neural pathways for colorectal control, relevance to spinal cord injury and treatment: a narrative review. Spinal Cord. 2018 Mar;56(3):199-205. doi: 10.1038/s41393-017-0026-2. Epub 2017 Nov 16. PMID 29142293
- [Result] Rao M, Gershon MD. The bowel and beyond: the enteric nervous system in neurological disorders. Nat Rev Gastroenterol Hepatol. 2016 Sep;13(9):517-28. doi: 10.1038/nrgastro.2016.107. Epub 2016 Jul 20. PMID 27435372
- [Result] Carabotti M, Scirocco A, Maselli MA, Severi C. The gut-brain axis: interactions between enteric microbiota, central and enteric nervous systems. Ann Gastroenterol. 2015 Apr-Jun;28(2):203-209. PMID 25830558
- [Result] Browning KN, Travagli RA. Central control of gastrointestinal motility. Curr Opin Endocrinol Diabetes Obes. 2019 Feb;26(1):11-16. doi: 10.1097/MED.0000000000000449. PMID 30418187
- [Result] Browning KN, Travagli RA. Central nervous system control of gastrointestinal motility and secretion and modulation of gastrointestinal functions. Compr Physiol. 2014 Oct;4(4):1339-68. doi: 10.1002/cphy.c130055. PMID 25428846
- [Result] Ali MK, Saha S, Milkova N, Liu L, Sharma K, Huizinga JD, Chen JH. Modulation of the autonomic nervous system by one session of spinal low-level laser therapy in patients with chronic colonic motility dysfunction. Front Neurosci. 2022 Sep 1;16:882602. doi: 10.3389/fnins.2022.882602. eCollection 2022. PMID 36117615
- [Result] Ali MK, Chen JDZ. Roles of Heart Rate Variability in Assessing Autonomic Nervous System in Functional Gastrointestinal Disorders: A Systematic Review. Diagnostics (Basel). 2023 Jan 12;13(2):293. doi: 10.3390/diagnostics13020293. PMID 36673103
- [Result] Yuan Y, Ali MK, Mathewson KJ, Sharma K, Faiyaz M, Tan W, Parsons SP, Zhang KK, Milkova N, Liu L, Ratcliffe E, Armstrong D, Schmidt LA, Chen JH, Huizinga JD. Associations Between Colonic Motor Patterns and Autonomic Nervous System Activity Assessed by High-Resolution Manometry and Concurrent Heart Rate Variability. Front Neurosci. 2020 Jan 23;13:1447. doi: 10.3389/fnins.2019.01447. eCollection 2019. PMID 32038145
- [Result] Ali MK, Liu L, Chen JH, Huizinga JD. Optimizing Autonomic Function Analysis via Heart Rate Variability Associated With Motor Activity of the Human Colon. Front Physiol. 2021 Jun 29;12:619722. doi: 10.3389/fphys.2021.619722. eCollection 2021. PMID 34267670
- [Result] Chen J. Neuromodulation and Neurostimulation for the Treatment of Functional Gastrointestinal Disorders. Gastroenterol Hepatol (N Y). 2022 Jan;18(1):47-49. No abstract available. PMID 35505768
- [Result] Yu Y, Wei R, Liu Z, Xu J, Xu C, Chen JDZ. Ameliorating Effects of Transcutaneous Electrical Acustimulation Combined With Deep Breathing Training on Refractory Gastroesophageal Reflux Disease Mediated via the Autonomic Pathway. Neuromodulation. 2019 Aug;22(6):751-757. doi: 10.1111/ner.13021. Epub 2019 Jul 26. PMID 31347247
- [Result] Huang WJ, Shu CH, Chou KT, Wang YF, Hsu YB, Ho CY, Lan MY. Evaluating the autonomic nervous system in patients with laryngopharyngeal reflux. Otolaryngol Head Neck Surg. 2013 Jun;148(6):997-1002. doi: 10.1177/0194599813482103. Epub 2013 Mar 21. PMID 23520070
- [Result] Ouyang H, Yin J, Wang Z, Pasricha PJ, Chen JD. Electroacupuncture accelerates gastric emptying in association with changes in vagal activity. Am J Physiol Gastrointest Liver Physiol. 2002 Feb;282(2):G390-6. doi: 10.1152/ajpgi.00272.2001. PMID 11804862
- [Result] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Result] Shaffer F, McCraty R, Zerr CL. A healthy heart is not a metronome: an integrative review of the heart's anatomy and heart rate variability. Front Psychol. 2014 Sep 30;5:1040. doi: 10.3389/fpsyg.2014.01040. eCollection 2014. PMID 25324790
- [Result] Ciccone AB, Siedlik JA, Wecht JM, Deckert JA, Nguyen ND, Weir JP. Reminder: RMSSD and SD1 are identical heart rate variability metrics. Muscle Nerve. 2017 Oct;56(4):674-678. doi: 10.1002/mus.25573. Epub 2017 Apr 8. PMID 28073153
- [Result] Bigger JT Jr, Albrecht P, Steinman RC, Rolnitzky LM, Fleiss JL, Cohen RJ. Comparison of time- and frequency domain-based measures of cardiac parasympathetic activity in Holter recordings after myocardial infarction. Am J Cardiol. 1989 Sep 1;64(8):536-8. doi: 10.1016/0002-9149(89)90436-0. No abstract available. PMID 2773799
- [Result] DeGiorgio CM, Miller P, Meymandi S, Chin A, Epps J, Gordon S, Gornbein J, Harper RM. RMSSD, a measure of vagus-mediated heart rate variability, is associated with risk factors for SUDEP: the SUDEP-7 Inventory. Epilepsy Behav. 2010 Sep;19(1):78-81. doi: 10.1016/j.yebeh.2010.06.011. Epub 2010 Jul 27. PMID 20667792
- [Result] Umetani K, Singer DH, McCraty R, Atkinson M. Twenty-four hour time domain heart rate variability and heart rate: relations to age and gender over nine decades. J Am Coll Cardiol. 1998 Mar 1;31(3):593-601. doi: 10.1016/s0735-1097(97)00554-8. PMID 9502641
- [Result] Otzenberger H, Gronfier C, Simon C, Charloux A, Ehrhart J, Piquard F, Brandenberger G. Dynamic heart rate variability: a tool for exploring sympathovagal balance continuously during sleep in men. Am J Physiol. 1998 Sep;275(3):H946-50. doi: 10.1152/ajpheart.1998.275.3.H946. PMID 9724299
- [Result] Karemaker JM. Counterpoint: respiratory sinus arrhythmia is due to the baroreflex mechanism. J Appl Physiol (1985). 2009 May;106(5):1742-3; discussion 1744. doi: 10.1152/japplphysiol.91107.2008a. No abstract available. PMID 19414625
- [Result] Kocjan J, Adamek M, Gzik-Zroska B, Czyzewski D, Rydel M. Network of breathing. Multifunctional role of the diaphragm: a review. Adv Respir Med. 2017;85(4):224-232. doi: 10.5603/ARM.2017.0037. PMID 28871591
- [Result] Stauss HM. Heart rate variability. Am J Physiol Regul Integr Comp Physiol. 2003 Nov;285(5):R927-31. doi: 10.1152/ajpregu.00452.2003. No abstract available. PMID 14557228
- [Result] Ambrosino N, Paggiaro PL, Macchi M, Filieri M, Toma G, Lombardi FA, Del Cesta F, Parlanti A, Loi AM, Baschieri L. A study of short-term effect of rehabilitative therapy in chronic obstructive pulmonary disease. Respiration. 1981;41(1):40-4. doi: 10.1159/000194357. PMID 7244391
- [Result] Montano N, Cogliati C, Porta A, Pagani M, Malliani A, Narkiewicz K, Abboud FM, Birkett C, Somers VK. Central vagotonic effects of atropine modulate spectral oscillations of sympathetic nerve activity. Circulation. 1998 Oct 6;98(14):1394-9. doi: 10.1161/01.cir.98.14.1394. PMID 9760293
- [Result] Bernardi L, Gabutti A, Porta C, Spicuzza L. Slow breathing reduces chemoreflex response to hypoxia and hypercapnia, and increases baroreflex sensitivity. J Hypertens. 2001 Dec;19(12):2221-9. doi: 10.1097/00004872-200112000-00016. PMID 11725167
- [Result] Yadlapati R, Gyawali CP, Pandolfino JE; CGIT GERD Consensus Conference Participants. AGA Clinical Practice Update on the Personalized Approach to the Evaluation and Management of GERD: Expert Review. Clin Gastroenterol Hepatol. 2022 May;20(5):984-994.e1. doi: 10.1016/j.cgh.2022.01.025. Epub 2022 Feb 2. Erratum In: Clin Gastroenterol Hepatol. 2022 Sep;20(9):2156. doi: 10.1016/j.cgh.2022.05.005. PMID 35123084
- [Result] Halland M, Bharucha AE, Crowell MD, Ravi K, Katzka DA. Effects of Diaphragmatic Breathing on the Pathophysiology and Treatment of Upright Gastroesophageal Reflux: A Randomized Controlled Trial. Am J Gastroenterol. 2021 Jan 1;116(1):86-94. doi: 10.14309/ajg.0000000000000913. PMID 33009052
- [Result] Naliboff BD, Benton D, Solomon GF, Morley JE, Fahey JL, Bloom ET, Makinodan T, Gilmore SL. Immunological changes in young and old adults during brief laboratory stress. Psychosom Med. 1991 Mar-Apr;53(2):121-32. doi: 10.1097/00006842-199103000-00002. PMID 2031066
- [Result] Jones R, Junghard O, Dent J, Vakil N, Halling K, Wernersson B, Lind T. Development of the GerdQ, a tool for the diagnosis and management of gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1030-8. doi: 10.1111/j.1365-2036.2009.04142.x. Epub 2009 Sep 8. PMID 19737151
- [Result] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Result] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Result] Revicki DA, Wood M, Wiklund I, Crawley J. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res. 1998 Jan;7(1):75-83. doi: 10.1023/a:1008841022998. PMID 9481153
- [Result] Taft TH, Triggs JR, Carlson DA, Guadagnoli L, Tomasino KN, Keefer L, Pandolfino JE. Validation of the oesophageal hypervigilance and anxiety scale for chronic oesophageal disease. Aliment Pharmacol Ther. 2018 May;47(9):1270-1277. doi: 10.1111/apt.14605. Epub 2018 Mar 12. PMID 29528128
- [Result] Lee Y, Yang MJ, Lai TJ, Chiu NM, Chau TT. Development of the Taiwanese Depression Questionnaire. Chang Gung Med J. 2000 Nov;23(11):688-94. PMID 11190378
- [Result] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Result] Taylor JM. Psychometric analysis of the Ten-Item Perceived Stress Scale. Psychol Assess. 2015 Mar;27(1):90-101. doi: 10.1037/a0038100. Epub 2014 Oct 27. PMID 25346996
- [Result] Labus JS, Bolus R, Chang L, Wiklund I, Naesdal J, Mayer EA, Naliboff BD. The Visceral Sensitivity Index: development and validation of a gastrointestinal symptom-specific anxiety scale. Aliment Pharmacol Ther. 2004 Jul 1;20(1):89-97. doi: 10.1111/j.1365-2036.2004.02007.x. PMID 15225175

DOCUMENTS (2):
  • Study Protocol (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT06205446/Prot_000.pdf
  • Informed Consent Form (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT06205446/ICF_001.pdf